CLINICAL TRIAL: NCT00690118
Title: Efficacy, Safety and Tolerability Study of 45 mg Pioglitazone in Patients With Amyotrophic Lateral Sclerosis (ALS) Receiving Standard Therapy (Riluzole)
Brief Title: Study of Pioglitazone in Patients With Amyotrophic Lateral Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The interim analysis showed no tendency in favour of the verum group. Therefore it was decided to stop the study prematurely.
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Albert Christian Ludolph, Prof., Coordinating Investigator, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GERP ALS; EUDRACT NUMBER 2006-005410-13
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; survival time; ALS functioning Rating Scale; quality of life; non-invasive ventilation; clinical tolerability; survival
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: pioglitazone
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pioglitazone — 45 mg/day, 18 months
  Other Names: Actos
  Arms: 1
Drug: placebo — once daily, 18 months
  Arms: 2

SUMMARY:
Primary objective:

Efficacy of pioglitazone (45 mg/day) as add-on therapy to standard therapy with riluzole in patients with ALS compared to placebo in terms of survival (mortality defined exclusively as death).

This is a prospective, multicentre, randomised, stratified, parallel-group, double-blind trial comparing placebo with 45 mg pioglitazone as add-on therapy to 100 mg riluzole in ALS in 220 enrolled patients. For entry, the El Escorial Criteria for diagnosis will be used. The duration of treatment will be 18 months. The primary endpoint will be subjected to a confirmatory analyses. Secondary variables will be incidence of tracheotomy or non-invasive ventilation, ALS Functional Rating Scale, Quality of life and safety variables.

ELIGIBILITY:
Inclusion Criteria:

* possible, probable (clinically or laboratory) or definite ALS according to the revised version of the El Escorial World Federation of Neurology criteria
* disease duration more than 6 months and less than 3 years
* best-sitting FVC between 50% and 95% of predicted normal
* continuously treated with 100 mg riluzole daily, for at least one month
* onset of progression weakness within 36 months prior to study
* women of childbearing age be non-lactating and surgically sterile or using a highly effective method of birth control and have a negative pregnancy test
* capable of thoroughly understanding all information given and giving full informed consent according to GCP

Exclusion Criteria:

* previous participation in another clinical study within the preceding three months
* tracheotomy or assisted ventilation of any type during the preceding three months
* gastrostomy
* any medical condition known to have an association with motor neuron dysfunction which might confound or obscure the diagnosis of ALS
* presence of any concomitant life-threatening disease or impairment likely to interfere with functional assessment
* confirmed hepatic insufficiency or abnormal liver function (ASAT and/or ALAT more than 1.5 upper limit of normal)
* renal insufficiency (serum creatinine more than 2.26 mg/dl)
* evidence of major psychiatric disorder or clinically evident dementia precluding evaluation of symptoms
* known hypersensitivity to any component of the study drugs
* likely to be not cooperative or comply with the trial requirements (as assessed by the investigator), or unable to be reached in the case of an emergency
* other antidiabetics
* heart failure or heart failure in the patients history (NYHA I to IV)
* history of macular oedema
* treatment with thiazolidinediones within 3 months prior to screening
* known or suspected history of alcohol and/or drug abuse
* treatment with gemfibrozil within 3 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2008-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Survival in patients with ALS treated with pioglitazone compared to placebo | 18 months

SECONDARY OUTCOMES:
Incidence of tracheotomy or non-invasive ventilation | 18 month

CONTACTS AND LOCATIONS:
Overall Officials: Albert C Ludolph, MD, Prof., Principal Investigator — Department of Neurology, University of Ulm
Locations (15):
- Germany (15):
  - Department of Neurology, University of Ulm, Ulm, Baden-Wurttemberg
  - Department of Neurology and Center for Palliative Medicine, University of Munich, Munich, Bavaria
  - Department of Neurology, Universty of Regensburg, Regensburg, Bavaria
  - Department of Neurology, University of Wuerzburg, Würzburg, Bavaria
  - Department of Neurology, Deutsche Klinik für Diagnostik, Wiesbaden, Hesse
  - Department of Neurology, University of Goettingen, Göttingen, Lower Saxony
  - Department of Neurology, Medical School Hannover, Hanover, Lower Saxony
  - Department of Neurology, University of Rostock, Rostock, Mecklenburg-Vorpommern
  - Department of Neurology, Universty of Bonn, Bonn, Nordrhrein-Westfalen
  - Neurologische Universitätsklinik Bergmannsheil, Bochum, North Rhine-Westphalia
  - Department of Neurology, Universty of Muenster, Münster, North Rhine-Westphalia
  - Department of Neurology, TU Dresden, Dresden, Saxony
  - Department of Neurology, University of Halle-Wittenberg, Halle, Saxony-Anhalt
  - Department of Neurology, University of Jena, Jena, Thuringia
  - Department of Neurology, Humboldt University, Berlin

REFERENCES:
- [Background] Schutz B, Reimann J, Dumitrescu-Ozimek L, Kappes-Horn K, Landreth GE, Schurmann B, Zimmer A, Heneka MT. The oral antidiabetic pioglitazone protects from neurodegeneration and amyotrophic lateral sclerosis-like symptoms in superoxide dismutase-G93A transgenic mice. J Neurosci. 2005 Aug 24;25(34):7805-12. doi: 10.1523/JNEUROSCI.2038-05.2005. PMID 16120782
- [Background] Kiaei M, Kipiani K, Chen J, Calingasan NY, Beal MF. Peroxisome proliferator-activated receptor-gamma agonist extends survival in transgenic mouse model of amyotrophic lateral sclerosis. Exp Neurol. 2005 Feb;191(2):331-6. doi: 10.1016/j.expneurol.2004.10.007. PMID 15649489
- [Derived] Dupuis L, Dengler R, Heneka MT, Meyer T, Zierz S, Kassubek J, Fischer W, Steiner F, Lindauer E, Otto M, Dreyhaupt J, Grehl T, Hermann A, Winkler AS, Bogdahn U, Benecke R, Schrank B, Wessig C, Grosskreutz J, Ludolph AC; GERP ALS Study Group. A randomized, double blind, placebo-controlled trial of pioglitazone in combination with riluzole in amyotrophic lateral sclerosis. PLoS One. 2012;7(6):e37885. doi: 10.1371/journal.pone.0037885. Epub 2012 Jun 8. PMID 22715372